CLINICAL TRIAL: NCT05663515
Title: EXCEED - A Pan-European Post-Authorisation Safety Study: Risk of Pancreatic Cancer Among Type 2 Diabetes Patients Who Initiated Exenatide as Compared With Those Who Initiated Other Non-Glucagon-Like Peptide 1 Receptor Agonists Based Glucose Lowering Drugs
Brief Title: A Pan-European Post-Authorisation Safety Study: Risk of Pancreatic Cancer Among Type 2 Diabetes Patients Who Initiated Exenatide as Compared With Those Who Initiated Other Non-Glucagon-Like Peptide 1 Receptor Agonists Based Glucose Lowering Drugs
Acronym: EXCEED
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: IQVIA Pvt. Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: D5551R00015
Record Dates: First submitted 2022-10-11; First posted 2022-12-23 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Exenatide; Insulin; Biguanides; Sulfonylurea Compounds; Sulfonamides; 2,4-thiazolidinedione

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

GROUPS / COHORTS (2):
- Initiators of exenatide: Patients with T2DM, aged 18 years or older, who initiated treatment with exenatide during the study period, 2006 to 2023
  Interventions: Drug: Exenatide
- Initiators of non-GLP-1 RA based glucose lowering drugs: Patients with T2DM, aged 18 years or older, who initiated treatment with non-GLP-1 RA based glucose lowering drugs during the study period, 2006 to 2023
  Interventions: Drug: Non-GLP-1 RA based glucose lowering drugs

INTERVENTIONS:
Drug: Exenatide — All patients initiating exenatide during the study period will be identified by ATC codes and be included in the exenatide group in a hierarchical manner, regardless of previous use of non-GLP-1 RA based glucose lowering drugs.
  Other Names: BYETTA, BYDUREON/BYDUREON BCise
  Groups: Initiators of exenatide
Drug: Non-GLP-1 RA based glucose lowering drugs — Initiators of non-GLP-1 RA based GLDs with no use of exenatide before or during the study period.
  Other Names: Insulin/analogues (excl. A10AE54, A10A56), Biguanide, Sulfonylurea, Sulfonamide (heterocycl.), combined oral GLD (excl. DPP-4i), Alpha glucose inhib., Thiazolidinedione, SGLT2i, Oth. GLD excl. insulin
  Groups: Initiators of non-GLP-1 RA based glucose lowering drugs

SUMMARY:
EXCEED is a non-interventional post-authorisation safety study aiming to assess the risk of developing pancreatic cancer among type 2 diabetes mellitus (T2DM) patients who initiated exenatide compared to those who initiated other non-glucagon like peptide 1 receptor agonists (GLP-1 RA) based glucose lowering drugs (GLDs). Study data will be collected from secondary data sources across 7 European countries. The study will be conducted as a multi-country, long-term, retrospective, observational database study. Initiators of exenatide will be matched to initiators of non-GLP-1 RA based GLDs (comparator group) based on propensity score and calendar period of study entry. All analyses for pancreatic cancer will be conducted in the matched study population using an "intention-to-treat" approach. The study will use information from 8 data sources in 7 European countries (France, Spain, The United Kingdom, Finland, Denmark, Norway, and Sweden). Patients with T2DM, aged 18 years or older, who initiated treatment with exenatide or non-GLP-1 RA based GLDs during the study period, 2006 to 2023, will be included. Exposure to exenatide and non-GLP-1 RA based GLDs will be ascertained from recordings of prescriptions or insurance claims registrations as available in the different data sources. The outcome of pancreatic cancer will be defined as a primary diagnosis of pancreatic cancer during follow-up.

ELIGIBILITY:
For inclusion in either exposure group, all of the following inclusion criteria must be fulfilled:

1. Aged 18 years or older at the index date
2. Individual level data on prescriptions, diagnoses and medical history is available for a minimum of 12 months prior to the index date
3. A diagnosis of T2DM on index date or prior to index date

For inclusion in the overall exenatide exposure group, the following criterion must be fulfilled:

1. One incident prescription (or incident dispensed prescription) for exenatide (BYETTA or BYDUREON/ BYDUREON BCise) between the start and 12 months before the end of the study period. This incident prescription must have succeeded a prescription of a GLD of another drug class during the baseline period.

   For inclusion in the BYDUREON/ BYDUREON BCise exposure group, for the analyses of the secondary objective, the criterion a) is substituted with criterion b):
2. One incident prescription (or incident dispensed prescription) for BYDUREON/ BYDUREON BCise between the start and 12 months before the end of the study period. This incident prescription must have succeeded a prescription of a GLD of another drug class during the baseline period.

   For inclusion in the comparator group, the following criterion must be fulfilled:
3. One incident prescription (or incident dispensed prescription) of a GLD between the start and 12 months before the end of the study period. The GLD must not be a DPP-4i, a GLP-1 RA, or a combination with either a DPP-4i or a GLP-1 RA. This incident prescription must have succeeded a prescription of a GLD of another drug class during the baseline period.

Patients are not eligible for any of the study population groups if they fulfil any of the following exclusion criteria:

1. A diagnosis of type 1 diabetes mellitus (T1DM) on index date or a diagnosis of T1DM during the baseline period that is not succeeded by a T2DM diagnosis during the remaining part of the baseline period.
2. A diagnosis of gestational diabetes during the baseline period or on index date.
3. A diagnosis of polycystic ovarian syndrome during the baseline period or on index date in combination with exposure to metformin (Anatomical Therapeutic Chemical Classification System (ATC) code of the World Health Organization (WHO): A10BA02) as the only GLD on index date or during the baseline period.
4. History of any cancer on or prior to index date. The only exception is that nonmelanoma skin cancer does not lead to exclusion.
5. History of any acute pancreatitis, other diseases of the pancreas, or disorders of the pancreas on or prior to index date.
6. One or more prescriptions (or dispensed prescriptions) of a GLP-1 RA (incretin mimetics) other than exenatide on or prior to index date.
7. One or more prescriptions (or dispensed prescriptions) of DPP-4i (incretin mimetics) on or prior to the index date.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with T2DM, aged 18 years or older, who initiated treatment with exenatide or non-GLP-1 RA based GLDs during the study period, 2006 to 2023, will be included. Exposure to exenatide and non-GLP-1 RA based GLDs will be ascertained from recordings of prescriptions or insurance claims registrations as available in the different data sources.
Sampling Method: Non-Probability Sample
Enrollment: 24000 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2026-03-02 (Estimated); Study Completion 2026-03-02 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of primary diagnosis of pancreatic cancer among exenatide exposed population | Follow-up starts from the index date to the study completion, an average of 1.5 years or less
  To estimate the incidence rate (IR) for pancreatic cancer associated with exposure to exenatide, compared with exposure to non-GLP-1 RA based GLDs, among patients with T2DM.
Hazard ratio of primary diagnosis of pancreatic cancer among exenatide exposed population | Follow-up starts from thr index date to the study completion, an average of 1.5 years or less
  To estimate the hazard ratio (HR) for pancreatic cancer associated with exposure to exenatide, compared with exposure to non-GLP-1 RA based GLDs, among patients with T2DM.

CONTACTS AND LOCATIONS:
Overall Officials: Fabian Hoti, PhD, Principal Investigator — Iqvia Pty Ltd
Locations (8):
- Research Site, Copenhagen, Denmark
- Research Site, Helsinki, Finland
- Research Site, Paris, France
- Research Site, Bergen, Norway
- Research Site, Barcelona, Spain
- Research Site, Vänersborg, Sweden
- United Kingdom (2):
  - Research Site, Edinburgh
  - Research Site, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/